CLINICAL TRIAL: NCT07349875
Title: Colchicine Treatment for Non-Flow-Limiting Coronary Plaque by Coronary CTA: A Randomized Controlled Trial
Acronym: COLOR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20241217-10-KS-02
Record Dates: First submitted 2025-12-29; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: Chronic coronary syndromes; Coronary Artery Disease (CAD); Coronary Artery Disease; COLCHICINE; Vulnerable Plaque
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guideline-Directed Medical Therapy Group (No Intervention): Guideline-directed medical therapy (GDMT) alone Guideline-directed medical therapy is based on the Guidelines for the Diagnosis and Management of Patients with Chronic Coronary Syndromes in China and includes the following types of drug therapies: antiplatelet drugs (aspirin, indobufen, or clopidogrel); anticoagulant drugs (warfarin or new oral anticoagulants); lipid-lowering drugs (control target: LDL-C < 1.8 mmol/L with a reduction of ≥50% from baseline; for ultra-high-risk patients, LDL-C < 1.4 mmol/L with a reduction of ≥50% from baseline); drugs for relieving symptoms such as β-blockers, nitrates, and calcium channel blockers. The specific drug selection and treatment plan will be adjusted according to the clinician's judgment and the actual situation of the patient.
- Colchicine plus Guideline-Directed Medical Therapy Group (Experimental): Guideline-directed medical therapy (GDMT) plus colchicine (0.5 mg once daily) Guideline-directed medical therapy is based on the Guidelines for the Diagnosis and Management of Patients with Chronic Coronary Syndromes in China and includes the following types of drug therapies: antiplatelet drugs (aspirin, indobufen, or clopidogrel); anticoagulant drugs (warfarin or new oral anticoagulants); lipid-lowering drugs (control target: LDL-C < 1.8 mmol/L with a reduction of ≥50% from baseline; for ultra-high-risk patients, LDL-C < 1.4 mmol/L with a reduction of ≥50% from baseline); drugs for relieving symptoms such as β-blockers, nitrates, and calcium channel blockers. The specific drug selection and treatment plan will be adjusted according to the clinician's judgment and the actual situation of the patient.
  Interventions: Drug: Colchicine combined with Guideline-Directed Medical Therapy

INTERVENTIONS:
Drug: Colchicine combined with Guideline-Directed Medical Therapy — colchicine combined with guideline-directed medical therapy group
  Arms: Colchicine plus Guideline-Directed Medical Therapy Group

SUMMARY:
This study is a prospective, multicenter, randomized controlled clinical trial designed to evaluate whether an anti-inflammatory medication can help improve heart health in patients with stable coronary artery disease.

1. Research Question & Hypothesis We aim to determine whether adding low-dose colchicine (0.5 mg once daily) to standard medical treatment can further reduce the risk of major cardiovascular events in patients with chronic coronary syndromes (CCS), especially those with non-flow-limiting coronary plaques detected by coronary CT angiography (CCTA).

   We hypothesize that colchicine, by reducing vascular inflammation, may help prevent future heart attacks, strokes, and the need for coronary revascularization.
2. Study Population & Design Design: A rigorously designed, prospective, multicenter, randomized (1:1), controlled superiority trial.

   Population: Adults (>18 years) diagnosed with CCS, identified by CCTA as having at least one coronary artery with ≥50% narrowing but without significant impact on blood flow (CT-FFR > 0.80).

   Intervention:

   Intervention Group: Standard guideline-directed medical therapy (GDMT) + colchicine 0.5 mg once daily Control Group: GDMT alone Sample Size: Approximately 3,826 participants, accounting for a 5% dropout rate.
3. Study Endpoints Primary Endpoint: The occurrence of major adverse cardiovascular or cerebrovascular events (MACCE), including:Cardiovascular death; Ischemic stroke; Non-fatal myocardial infarction; Any coronary revascularization. Assessed for 12 months after the last patient is enrolled.

Secondary Endpoints:Occurrence of MACCE over 36 months. Incidence and time to first occurrence of each event category at 12, 24, and 36 months.

Safety Endpoint: Side effects related to colchicine (e.g., gastrointestinal upset, liver or kidney abnormalities, blood disorders, muscle-related reactions).

ELIGIBILITY:
Inclusion Criteria

1. The subject (or legal guardian) understands the trial requirements and treatment procedure, and signs the written informed consent before undergoing any protocol-specified examinations or procedures;
2. Aged ≥18 years;
3. Clinically diagnosed with chronic coronary syndrome (CCS);
4. CCTA confirms ≥50% stenosis in at least one epicardial coronary artery, and CT fractional flow reserve (CT-FFR) >0.80.

Exclusion Criteria

1. Unable or unwilling to provide informed consent;
2. Unable to complete scheduled follow-up;
3. Underwent PCI within the past 3 months;
4. History of coronary artery bypass grafting (CABG);
5. Diagnosis of acute coronary syndromes (ACS);
6. No coronary plaque or plaque stenosis <50% (confirmed by CCTA);
7. Lesion-specific CT-FFR ≤0.80 in at least one major epicardial coronary artery;
8. Inflammatory bowel disease (Crohn's disease/ulcerative colitis) or chronic diarrhea;
9. History of gastric ulcer or gastric bleeding;
10. Pregnant/lactating women or women of childbearing age without effective contraception;
11. Neuromuscular disease or non-transient creatine kinase (CK) >3×upper limit of normal (ULN) (confirmed by ≥2 lab tests);
12. Clinically significant non-transient hematological abnormalities (hemoglobin <100 g/L, hematocrit <30%/ >52%, white blood cell count <3×10⁹/L, platelet count <100×10⁹/L; confirmed by ≥2 lab tests);
13. Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m² (CKD-EPI formula);
14. Liver dysfunction (alanine aminotransferase >3×ULN and/or total bilirubin >2×ULN);
15. Current/planned immunosuppressive therapy;
16. Long-term colchicine use for other indications;
17. Definite/suspected colchicine allergy;
18. Active malignant tumor (expected survival <1 year);
19. Use of potent CYP3A4/P-glycoprotein inhibitors (e.g., cyclosporine, antiretrovirals, antifungals, erythromycin, clarithromycin) without alternative drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3826 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2029-12-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular and cerebrovascular events (MACCE) | 12 months after enrollment
  Composite of cardiovascular death, ischemic stroke, non-fatal myocardial infarction, and any coronary revascularization (follow-up ends when the last enrolled patient completes 12 months of follow-up).

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, China

IPD SHARING:
Plan to Share IPD: No